CLINICAL TRIAL: NCT01350440
Title: Safety and Efficacy of Intravenous Immune Globulin in Treating Spinocerebellar Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Theresa Zesiewicz, Professor of Neurology, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2011-04-20; First posted 2011-05-09 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Spinocerebellar Ataxia
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Immunoglobulins, Intravenous

ARMS (1):
- IVIG (Experimental): Intravenous Immune Globulin
  Interventions: Biological: IVIG

INTERVENTIONS:
Biological: IVIG — Intravenous Immune Globulin

SUMMARY:
This is a preliminary study to determine the safety and efficacy of intravenous immune globulin in treating Spinocerebellar Ataxia. The investigators aim to assess changes in clinical measures of disease severity before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with SCA diagnosed by a movement disorder specialist.
2. Age 10 years to 80 years.
3. Able to ambulate with or without assistance for 30 feet.
4. Women of child-bearing potential must use a reliable method of contraception and must provide a negative pregnancy test at entry into the study.
5. Serum creatine kinase, complete metabolic panel, complete blood count, liver function tests, renal function tests, platelets and EKG do not reveal clinically significant abnormalities (results obtained from primary care physician and dated within the past 6 months or obtained at screening visit).
6. Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
7. Stable doses of all antidepressants and vitamins (including internet purchased idebenone) for 30 days prior to study entry and for the duration of the study. Throughout the study, all possible efforts should be made to maintain stable doses of all other medications.
8. Subject permission (informed consent).

Exclusion Criteria:

1. Any unstable illness that in the investigator's opinion precludes participation in this study.
2. Use of any investigational product within the past 30 days.
3. Presence of clinically significant cardiac disease (as determined by the investigator based on EKG and echocardiogram results within the past 6 months). Specifically, an ejection fraction <40%, or a prolonged QT interval (>50% of cycle duration) will be excluded. If the investigator notes clinically significant abnormalities on the EKG or echocardiogram, the subject will be eligible IF they provide clearance from a cardiologist.
4. Presence of diabetes (as determined by blood glucose labs within the past 6 months).
5. Dementia or other psychiatric illness that prevents the subject from giving informed consent (MMSE less than 25).
6. Legal incapacity or limited legal capacity.
7. Presence of severe renal disease (estimated creatinine clearance <50 mL/min) or hepatic disease (AST or ALT>2x times normal) (as evidenced by labs reported within the past 6 months).
8. Clinically significantly abnormal WBC, hemoglobin or platelet count (as evidenced by labs reported within the past 6 months).
9. IgA deficiency (evidenced by screening lab evaluations)

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia | participants will be followed for approximately 4 months

SECONDARY OUTCOMES:
Timed 25 foot walk | participants will be followed for approximately 4 months
Clinical Global impression | participants will be followed for approximately 4 months
Biodex Balance SD | participants will be followed for approximately 4 months
Gait Rite Mat | participants will be followed for approximately 4 months
Berg balance scale | participants will be followed for approximately 4 months
Complete Metabolic Panel | participants will be followed for approximately 4 months
Complete Blood Count | participants will be followed for approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States